CLINICAL TRIAL: NCT03570099
Title: Naloxone Treatment in Skåne County - Effect on Drug-related Mortality and Overdose-related Complications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/300
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Opioid Abuse
Keywords: opioid overdose; mortality; naloxone; substance use disorder; prevention
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Naloxone cohort: The prospective cohort consists of study subjects receiving Naloxone nasal spray in the distribution program.
  Interventions: Drug: Naloxone Nasal Spray
- Historical control cohort: Data from the historical control cohort will be collected from national registries years 2013-2017.
  Interventions: Other: Historical control cohort

INTERVENTIONS:
Drug: Naloxone Nasal Spray — Naloxone Nasal Spray will be distributed at the addiction centres.
  Groups: Prospective Naloxone cohort
Other: Historical control cohort — Historical data will be retrieved from quality registries.
  Groups: Historical control cohort

SUMMARY:
Death in overdose is the single most common cause of death in people using heroin. In Sweden, the number of drug-related overdose deaths has increased gradually since the early 1990s. The purpose of the study is to investigate the effects of a Naloxone distribution program in Skåne County. The primary issue is whether the project had an effect on overdose mortality and overdose related injuries.

ELIGIBILITY:
Inclusion Criteria:

* subjects treated at the Addiction centres of Skåne County
* signed informed consent

Exclusion Criteria:

* subjects unable to understand study information due to psychiatric co-morbidity or severe language difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects treated at the Addiction centres of Skåne County. Naloxone Nasal Spray will be handed out to these subjects, who must be able to understand the given information about the use of the drug.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Overdose mortality in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Overdose mortality deaths 2019-2023 to be compared with historical overdose mortality during 2013-2017. Number of deaths will be collected from national registries.

SECONDARY OUTCOMES:
Reaction level of ambulance-attended opioid overdose survivors in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Assessment of responsiveness in acute brain disorders using Reaction Level Scale (RLS-85) in ambulance. The RLS scale is graded from 1 (awake, no delayed reaction, oriented) to grade 8 (unconscious, no movements to painful stimuli).
Respiratory rate of ambulance-attended opioid overdose survivors in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Respiratory rate (breaths per minute) registered in ambulance.
Heart rate of ambulance-attended opioid overdose survivors in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Heart rate (beats per minute) of opioid overdose survivors registered in ambulance.
Naloxone or other antidot administered by ambulance staff to ambulance-attended opioid overdose survivors in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Naloxone or other antidot, if needed, administered by ambulance staff in opioid overdose survivors.
Need of ambulance transport to hospital of ambulance-attended opioid overdose survivors in the general population | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  The need to transport the opioid overdose survivors to hospital - information registered in ambulance.
Incidence of opioid overdoses attended by ambulance or emergency hospital care | 5 years (first outcome measure for the 18-month intervention period July 1, 2019 - Dec 31, 2020)
  Incidence of opioid overdoses attended by ambulance or emergency hospital care, information registered in ambulance or emergency hospital care.
All cause mortality in included patients | 3 years
  Number of deaths will be collected from national and regional registries.
Overdose mortality in included patients | 3 years
  Overdose mortality in included patients. Number of deaths will be collected from national and regional registries.
Retention in naloxone program | 3 years
  Retention in naloxone program - number of patients.
Incidence of witnessing opioid overdoses | 3 years
  Number of incidences of witnessing opioid overdoses.
Incidence in naloxone use and bystander CPR | 3 years
  Number of incidences of naloxone use and bystander CPR.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmqvist, MD, PhD, Study Director — Region Skåne
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Troberg K, Isendahl P, Dahlman D, Hakansson A. Broad-scale overdose education and naloxone distribution- 5-year follow-up of a regional program in Skane County, Sweden. Harm Reduct J. 2025 Jun 5;22(1):97. doi: 10.1186/s12954-025-01255-3. PMID 40474253
- [Derived] Hakansson A, Alanko Blome M, Isendahl P, Landgren M, Malmqvist U, Troberg K. Distribution of intranasal naloxone to potential opioid overdose bystanders in Sweden: effects on overdose mortality in a full region-wide study. BMJ Open. 2024 Jan 3;14(1):e074152. doi: 10.1136/bmjopen-2023-074152. PMID 38171623
- [Derived] Troberg K, Isendahl P, Blome MA, Dahlman D, Hakansson A. Protocol for a multi-site study of the effects of overdose prevention education with naloxone distribution program in Skane County, Sweden. BMC Psychiatry. 2020 Feb 7;20(1):49. doi: 10.1186/s12888-020-2470-3. PMID 32028921